CLINICAL TRIAL: NCT03727659
Title: CONNECT: A Social Media Intervention for Depressed Cannabis Users
Brief Title: CONNECT for Depressed Cannabis Users Trial
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Suzette Glasner-Edwards, Research Psychologist, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT
Record Dates: First submitted 2018-10-17; First posted 2018-11-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Substance Abuse; Depression
Keywords: Cannabis; CONNECT; Depression; FaceBook
MeSH Terms: conditions — Substance-Related Disorders; Depression; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Participants will receive SHADE therapy for drug use and depression for 10 weeks plus CONNECT FaceBook social support.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHADE therapy + CONNECT FaceBook support (Experimental): SHADE is a 10-week, 10-session, computerized CBT/MET intervention for Cannabis Use Disorder and depression. At each visit, a study clinician meets with participants for a 'check-in' session, which includes: review of homework; plans for completing homework; suicide risk and mood assessment. The CONNECT FB intervention component will facilitate social support for between-session homework and CBT skills practice for managing depression and preventing relapse, and bolstering motivation to change. Daily posts will be delivered. Only those participating in the study will know about the existence of this group and will be able to access it. A weekly real-time, Facebook chat session will be held to provide feedback concerning homework practice or answer questions.
  Interventions: Behavioral: SHADE therapy + CONNECT FaceBook support

INTERVENTIONS:
Behavioral: SHADE therapy + CONNECT FaceBook support — See "study arms" description.

SUMMARY:
The purpose of this study is to test the usefulness of a computer-assisted intervention for depressed cannabis users by combining peer and therapist social network support via Facebook that uses the techniques of cognitive behavioral therapy and motivational enhancement therapy (CBT/MET) to help with relapse prevention skills, reduce cannabis use and depressive symptoms, and improve treatment adherence. All participants will receive 10 weeks of the computer assisted intervention which includes weekly 60 minute (1 hour) sessions. All participants will also be part of a secret Facebook group (CONNECT). The goal of this secret Facebook group is to reinforce the knowledge and skills taught in the computer assisted intervention and to provide social support.

DETAILED DESCRIPTION:
An estimated 8.4 million adults in the U.S. experience co-occurring psychiatric and SUDs, largely accounted for by comorbid mood disorder-SUD. Cannabis is the most widely used illicit substance among individuals with depressive disorders1. Likewise, elevated rates of major depression are observed among those with cannabis use disorders (CUD)2.

The use of technology-based platforms for behavioral intervention delivery in primary care settings, focusing on comorbidity, is a promising approach to broadening availability of evidence-based treatments for this high-need population, at low cost.

With support from a NIDA High Priority, Short-Term Project Award, the present investigative team (PI Dr. Glasner-Edwards and Drs. Budney and Kay-Lambkin) piloted SHADE (Self-Help for Alcohol and Other Drug Use and Depression), a computerized intervention model combining cognitive behavioral therapy (CBT) and motivational enhancement therapy (MET), in a primary psychiatric care setting, where integrated interventions addressing both mental health and SUDs are not readily accessible. Preliminary data indicate that SHADE: (1) was feasible and acceptable, (2) facilitated treatment engagement and retention in a difficult-to-treat comorbid population with major depression and CUD; and (3) effectively reduced cannabis use and depression. As a next step to optimize the efficacy of this intervention model, the present proposal is designed to develop and integrate a social media component to the SHADE intervention program, based on a program established and tested by Co-I Dr. Ramo in an RCT4.

To this end, we propose to: (a) develop and refine, with user feedback, a social media-assisted therapy intervention, CONNECT (Connected Cannabis Users' Network for Enhancement of Cognitive Therapy), which combines the use of Facebook for social network support with SHADE in a population of adults with CUD and major depression; and (b) collect preliminary data to evaluate effect sizes and investigate trends for the impact of CONNECT plus SHADE on cannabis use, depressive symptoms, and health service utilization. Moreover, we will gather preliminary data for social network analysis, to understand the mechanism(s) by which the social media component of CONNECT promotes health behavior change in the key outcome domains of the present study.

The use of a social media platform (i.e., Facebook) will increase the accessibility of the intervention as Facebook can be accessed using a variety of technology devices.

Aim 1. To develop and refine, with user feedback, a 10-week, social media-assisted intervention (CONNECT) combining a computer-assisted, integrated treatment program (SHADE) with private Facebook groups to facilitate peer and clinician support for therapeutic objectives. The CONNECT intervention targets cannabis use and depression in a population of depressed adults with CUD receiving psychiatric care.

Hypothesis 1: Participants will report that CONNECT is user-friendly and helpful in providing opportunities for between-session practice of therapy skills, peer and clinician support, and information that enable them to prevent cannabis relapse and manage depression.

Aim 2. To test the impact of CONNECT plus SHADE on cannabis use, depression, adherence to psychiatric care, and healthcare outcomes.

Hypothesis 2a: Among depressed substance dependent adults in an outpatient psychiatric care setting, CONNECT plus SHADE will led to clinical outcomes in reducing cannabis use and depression, and improving adherence to psychiatric care during and after treatment.

Aim 3. To test whether social network variables mediate or moderate the impact of CONNECT.

Hypothesis 3: Participants with more expansive Facebook social networks within CONNECT will benefit more from the program. Factors that influence engagement in the Facebook component of CONNECT will also be explored (e.g., social network characteristics and content of peer and therapist interaction via the social network), and engagement will be examined as a potential moderator of cannabis use and depression outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 65;
2. DSM-5 diagnosis of CUD, with use reported on >50 of the past 90 days;
3. DSM-5 diagnosis of Major Depressive Disorder (Lifetime);
4. Current Patient Health Questionnaire-9 (PHQ9) score > 9;
5. Uses Facebook or willing to join and learn how to use it;
6. Having received treatment for depression in the past year.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in illicit drug use between study visits and at follow up | Baseline (week 0), weekly during treatment (weeks 1-10), and follow up (week 14).
  Substance use will be tracked with urine drug screens between each study visit.
Change in depression symptoms and severity between study visits and at follow up | Baseline (week 0), weekly during treatment (weeks 1-10) and follow up (week 14)
  Depression will be tracked with a questionnaire designed to capture frequency and severity of depression symptoms; Patient Health Questionnaire-9 (PHQ9) at each study visit. The scale of the PHQ-9 is 0-27 where 0-4=Minimal or none; 5-9=Mild; 10-14=Moderate; 15-19=Moderately severe; 20-27=Severe.
Change in adherence to collateral psychiatric treatment between study visits and at follow up | Baseline (week 0), weekly during treatment (weeks 1-10), and follow up (week 14)
  Treatment adherence to collateral therapy and medication will be tracked with self-report questionnaire (Ancillary Treatment Record).

SECONDARY OUTCOMES:
Change in alcohol use between study visits and at follow up | Baseline (week 0), weekly during treatment (weeks 1-10), and follow up (week 14)
  Breathalyzer test will be used at each study visit to obtain blood alcohol level.
Change in alcohol, tobacco and other drug use between study visits and at follow up | Baseline (week 0), weekly during treatment (weeks 1-10), and follow up (week 14)
  Alcohol tobacco and other drug use will be obtained through verbal history using the Timeline follow back (TLFB) interview at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Glasner, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Integrated Substance Abuse Programs, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Background] Glasner-Edwards S, Rawson R. Evidence-based practices in addiction treatment: review and recommendations for public policy. Health Policy. 2010 Oct;97(2-3):93-104. doi: 10.1016/j.healthpol.2010.05.013. Epub 2010 Jun 16. PMID 20557970
- [Background] Aspis I, Feingold D, Weiser M, Rehm J, Shoval G, Lev-Ran S. Cannabis use and mental health-related quality of life among individuals with depressive disorders. Psychiatry Res. 2015 Dec 15;230(2):341-9. doi: 10.1016/j.psychres.2015.09.014. Epub 2015 Sep 10. PMID 26388103
- [Background] Cornelius JB, Cato MG, Toth JL, Bard PM, Moore MW, White A. Following the trail of an HIV-prevention Web site enhanced for mobile cell phone text messaging delivery. J Assoc Nurses AIDS Care. 2012 May-Jun;23(3):255-9. doi: 10.1016/j.jana.2011.03.002. Epub 2011 May 7. No abstract available. PMID 21550826